CLINICAL TRIAL: NCT05757167
Title: Improving Neonatal Health Through Rapid Malaria Testing in Early Pregnancy With High-Sensitivity
Brief Title: Improving Neonatal Health Through Rapid Malaria Testing in Early Pregnancy With High-Sensitivity Diagnostics
Acronym: INTREPiD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Pro00110771; 1U01AI162463-01A1 (NIH); 5U01AI162463-02 (NIH); 5U01AI162463-03 (NIH); 5U01AI162463-04 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malaria,Falciparum; Malaria in Pregnancy; Malaria in Childbirth; Pregnancy; Neonatal Health; Low Birthweight; Stillbirth; Gestational Age and Weight Conditions; Preterm Birth
MeSH Terms: conditions — Malaria, Falciparum; Stillbirth; Premature Birth | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Random assignment to either a) usual antenatal care or b) testing for malaria with a high-sensitivity rapid diagnostic test followed by treatment with artemether-lumefantrine if tested positive
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HS-RDT screening/AL treatment (Experimental): Pregnant women will be screened with a malaria HS-RDT and, if positive, treated with artemether-lumefantrine
  Interventions: Diagnostic Test: Malaria High-Sensitivity Rapid Diagnostic Test (HS-RDT); Drug: Artemether-lumefantrine (AL)
- Usual antenatal care (No Intervention): Pregnant women will receive usual antenatal care

INTERVENTIONS:
Diagnostic Test: Malaria High-Sensitivity Rapid Diagnostic Test (HS-RDT) — Detection of Plasmodium falciparum HRP-II antigen1
  Method: Lateral Flow; Time to Result: 20 minutes; Sample Type: Fingerstick Whole Blood; Sample Volume: 5µl; Storage Conditions: 1-30°C; Shelf Life: 12 months; Sensitivity/Specificity: 99.0%/98.6%
  Other Names: NxTek™ Eliminate Malaria P.f; 05FK140 (Global); 05FK141 (Global); 05FK142 (Global); 05FK143 (Global); Alere Malaria Ag P.f
  Arms: HS-RDT screening/AL treatment
Drug: Artemether-lumefantrine (AL) — oral tablets: 6 doses of 80/480 mg over 3 days
  Other Names: AL
  Arms: HS-RDT screening/AL treatment

SUMMARY:
The purpose of the INTREPiD study is to compare 1st trimester screening for malaria parasites with a high-sensitivity malaria rapid diagnostic test followed by treatment of test-positive women with artemether-lumefantrine (AL) against usual antenatal care on a composite adverse pregnancy outcome including low birth weight, small for gestational age, preterm, fetal loss, or neonatal death.

DETAILED DESCRIPTION:
INTREPiD is a two-arm, open-label, parallel-assignment randomized trial of a strategy of 1st trimester screening for P. falciparum parasites with a high-sensitivity rapid diagnostic test (HS-RDT). Participants will be women of all gravidities presenting to antenatal clinics in the 1st trimester in sites endemic for P. falciparum malaria in Kenya and the Democratic Republic of the Congo.

Following consent and enrollment, women will be allocated 1:1 to either usual antenatal care or to the intervention. The intervention will be a single screening in the 1st trimester for P. falciparum infection in maternal peripheral blood with a HS-RDT. Women who test positive for P. falciparum on HS-RDT testing will be treated with a single course of Artemether-Lumefantrine (AL) and then returned to usual antenatal care.

Participants will be followed through delivery and then through their offspring's first month of life.

The Hypothesis is that, compared to usual antenatal care, screening women in the 1st trimester for P. falciparum and treating them if positive with AL will reduce the risk of an adverse pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 years and 40 years (inclusive)
* Viable singleton pregnancy with gestational age estimated less than 13 6/7 weeks (inclusive) by ultrasound
* HIV-uninfected
* Willing to participate in the study schedule
* Planning to remain in the study area for the duration of pregnancy and 1 month after delivery
* Willing to deliver in a study-affiliated health facility

Exclusion Criteria:

* High risk pregnancy that requires referral for specialized care by local guidelines
* Active medical problem at the time of screening requiring higher level care
* Antimalarial receipt in the 2 weeks prior to screening
* Past allergy to Artemether or Lumefantrine or another condition that prohibits the receipt of either drug
* Current participation in another clinical research study

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Composite number of adverse pregnancy outcomes | Enrollment to 28 days Post-delivery (including each antenatal care visit)
  Adverse pregnancy outcomes defined as low birth weight (<2500 grams) OR preterm (< 37 0/7 weeks) OR small for gestational age (GA) (< 10th percentile weight for GA) OR pregnancy loss, defined as a. spontaneous abortion ( loss < 22 0/7 weeks gestation) OR b. stillbirth (loss ≥ 22 0/7 weeks gestation) OR neonatal death (livebirth with death prior to the 28th day of life).

SECONDARY OUTCOMES:
Birthweight | Delivery
  Birthweight in grams
Number of infants with low birthweight | Delivery
  < 2500 grams, livebirth
Gestational age (GA) | Delivery
  GA at delivery in weeks/days, livebirth
Preterm | Delivery
  < 37 0/7 weeks, livebirth
Number of infants that are small for gestational age | Delivery
  Weight for gestational age < 10th percentile, livebirth
Number of adverse newborn outcomes | Delivery
  low birthweight OR preterm OR small for gestational age
Number of spontaneous abortions | Delivery
  Pregnancy loss < 22 0/7 weeks gestation
Number of stillbirths | Delivery
  Pregnancy loss ≥ 22 0/7 weeks gestation
Number of early fetal deaths | Delivery
  Pregnancy loss 22 0/7 - 27 6/7 weeks gestation
Number of late fetal deaths | Delivery
  Pregnancy loss ≥ 28 0/7 weeks gestation
Number of pregnancy losses | Delivery
  Spontaneous abortion OR stillbirth
Number of neonatal deaths | Delivery to 28 days Post-delivery
  Before the 28th day of life, livebirth
Number of perinatal deaths | Delivery to 28 days Post-delivery
  Late fetal death OR Neonatal death
Incidence of clinical malaria during pregnancy | Enrollment to Delivery (including each antenatal care visit)
  Maternal symptoms with peripheral malaria parasitemia detected by light microscopy or rapid diagnostic test
Number of mothers with peripheral parasitemia at delivery | Delivery
  Maternal peripheral parasitemia at delivery by PCR
Mean maternal hemoglobin concentration | Enrollment and Delivery
  Maternal hemoglobin (g/dL)
Number of mothers with anemia at delivery | Delivery
  Maternal Hb concentration ≤ 11 g/dL
Number of mothers with severe anemia at delivery | Delivery
  Maternal Hb concentration ≤ 7 g/dL

OTHER OUTCOMES:
Number of maternal serious adverse events | Enrollment to 28 days Post-delivery
  Serious adverse events in the mothers
Number of infants with congenital malformations | Delivery to 28 days Post-delivery
  Congenital malformations identified within the first 28 days of birth
Number of offspring with the need for hospitalization or acute medical evaluation | Delivery to 28 days Post-delivery
  Hospitalization or acute medical evaluation within the first 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Steve M Taylor, MD, MPH, Principal Investigator — Duke University
Locations (2):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Background] Rogerson SJ, Desai M, Mayor A, Sicuri E, Taylor SM, van Eijk AM. Burden, pathology, and costs of malaria in pregnancy: new developments for an old problem. Lancet Infect Dis. 2018 Apr;18(4):e107-e118. doi: 10.1016/S1473-3099(18)30066-5. Epub 2018 Jan 31. PMID 29396010
- [Background] Lawn JE, Blencowe H, Waiswa P, Amouzou A, Mathers C, Hogan D, Flenady V, Froen JF, Qureshi ZU, Calderwood C, Shiekh S, Jassir FB, You D, McClure EM, Mathai M, Cousens S; Lancet Ending Preventable Stillbirths Series study group; Lancet Stillbirth Epidemiology investigator group. Stillbirths: rates, risk factors, and acceleration towards 2030. Lancet. 2016 Feb 6;387(10018):587-603. doi: 10.1016/S0140-6736(15)00837-5. Epub 2016 Jan 19. PMID 26794078
- [Background] van Eijk AM, Larsen DA, Kayentao K, Koshy G, Slaughter DEC, Roper C, Okell LC, Desai M, Gutman J, Khairallah C, Rogerson SJ, Hopkins Sibley C, Meshnick SR, Taylor SM, Ter Kuile FO. Effect of Plasmodium falciparum sulfadoxine-pyrimethamine resistance on the effectiveness of intermittent preventive therapy for malaria in pregnancy in Africa: a systematic review and meta-analysis. Lancet Infect Dis. 2019 May;19(5):546-556. doi: 10.1016/S1473-3099(18)30732-1. Epub 2019 Mar 25. PMID 30922818
- [Background] Gonzalez R, Mombo-Ngoma G, Ouedraogo S, Kakolwa MA, Abdulla S, Accrombessi M, Aponte JJ, Akerey-Diop D, Basra A, Briand V, Capan M, Cot M, Kabanywanyi AM, Kleine C, Kremsner PG, Macete E, Mackanga JR, Massougbodgi A, Mayor A, Nhacolo A, Pahlavan G, Ramharter M, Ruperez M, Sevene E, Vala A, Zoleko-Manego R, Menendez C. Intermittent preventive treatment of malaria in pregnancy with mefloquine in HIV-negative women: a multicentre randomized controlled trial. PLoS Med. 2014 Sep 23;11(9):e1001733. doi: 10.1371/journal.pmed.1001733. eCollection 2014 Sep. PMID 25247709
- [Background] Divala TH, Mungwira RG, Mawindo PM, Nyirenda OM, Kanjala M, Ndaferankhande M, Tsirizani LE, Masonga R, Muwalo F, Boudova S, Potter GE, Kennedy J, Goswami J, Wylie BJ, Muehlenbachs A, Ndovie L, Mvula P, Mbilizi Y, Tomoka T, Laufer MK. Chloroquine as weekly chemoprophylaxis or intermittent treatment to prevent malaria in pregnancy in Malawi: a randomised controlled trial. Lancet Infect Dis. 2018 Oct;18(10):1097-1107. doi: 10.1016/S1473-3099(18)30415-8. Epub 2018 Sep 5. PMID 30195996
- [Background] Kimani J, Phiri K, Kamiza S, Duparc S, Ayoub A, Rojo R, Robbins J, Orrico R, Vandenbroucke P. Efficacy and Safety of Azithromycin-Chloroquine versus Sulfadoxine-Pyrimethamine for Intermittent Preventive Treatment of Plasmodium falciparum Malaria Infection in Pregnant Women in Africa: An Open-Label, Randomized Trial. PLoS One. 2016 Jun 21;11(6):e0157045. doi: 10.1371/journal.pone.0157045. eCollection 2016. PMID 27326859
- [Background] Tagbor H, Bruce J, Agbo M, Greenwood B, Chandramohan D. Intermittent screening and treatment versus intermittent preventive treatment of malaria in pregnancy: a randomised controlled non-inferiority trial. PLoS One. 2010 Dec 28;5(12):e14425. doi: 10.1371/journal.pone.0014425. PMID 21203389
- [Background] Madanitsa M, Kalilani L, Mwapasa V, van Eijk AM, Khairallah C, Ali D, Pace C, Smedley J, Thwai KL, Levitt B, Wang D, Kang'ombe A, Faragher B, Taylor SM, Meshnick S, Ter Kuile FO. Scheduled Intermittent Screening with Rapid Diagnostic Tests and Treatment with Dihydroartemisinin-Piperaquine versus Intermittent Preventive Therapy with Sulfadoxine-Pyrimethamine for Malaria in Pregnancy in Malawi: An Open-Label Randomized Controlled Trial. PLoS Med. 2016 Sep 13;13(9):e1002124. doi: 10.1371/journal.pmed.1002124. eCollection 2016 Sep. PMID 27622558
- [Background] Desai M, Gutman J, L'lanziva A, Otieno K, Juma E, Kariuki S, Ouma P, Were V, Laserson K, Katana A, Williamson J, ter Kuile FO. Intermittent screening and treatment or intermittent preventive treatment with dihydroartemisinin-piperaquine versus intermittent preventive treatment with sulfadoxine-pyrimethamine for the control of malaria during pregnancy in western Kenya: an open-label, three-group, randomised controlled superiority trial. Lancet. 2015 Dec 19;386(10012):2507-19. doi: 10.1016/S0140-6736(15)00310-4. Epub 2015 Sep 28. PMID 26429700
- [Background] Kajubi R, Ochieng T, Kakuru A, Jagannathan P, Nakalembe M, Ruel T, Opira B, Ochokoru H, Ategeka J, Nayebare P, Clark TD, Havlir DV, Kamya MR, Dorsey G. Monthly sulfadoxine-pyrimethamine versus dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria in pregnancy: a double-blind, randomised, controlled, superiority trial. Lancet. 2019 Apr 6;393(10179):1428-1439. doi: 10.1016/S0140-6736(18)32224-4. Epub 2019 Mar 22. PMID 30910321
- [Background] Kakuru A, Jagannathan P, Muhindo MK, Natureeba P, Awori P, Nakalembe M, Opira B, Olwoch P, Ategeka J, Nayebare P, Clark TD, Feeney ME, Charlebois ED, Rizzuto G, Muehlenbachs A, Havlir DV, Kamya MR, Dorsey G. Dihydroartemisinin-Piperaquine for the Prevention of Malaria in Pregnancy. N Engl J Med. 2016 Mar 10;374(10):928-39. doi: 10.1056/NEJMoa1509150. PMID 26962728
- [Background] Desai M, Gutman J, Taylor SM, Wiegand RE, Khairallah C, Kayentao K, Ouma P, Coulibaly SO, Kalilani L, Mace KE, Arinaitwe E, Mathanga DP, Doumbo O, Otieno K, Edgar D, Chaluluka E, Kamuliwo M, Ades V, Skarbinski J, Shi YP, Magnussen P, Meshnick S, Ter Kuile FO. Impact of Sulfadoxine-Pyrimethamine Resistance on Effectiveness of Intermittent Preventive Therapy for Malaria in Pregnancy at Clearing Infections and Preventing Low Birth Weight. Clin Infect Dis. 2016 Feb 1;62(3):323-333. doi: 10.1093/cid/civ881. Epub 2015 Oct 20. PMID 26486699
- [Background] Leuba SI, Westreich D, Bose CL, Powers KA, Olshan A, Taylor SM, Tshefu A, Lokangaka A, Carlo WA, Chomba E, Liechty EA, Bucher SL, Esamai F, Jessani S, Saleem S, Goldenberg RL, Moore J, Nolen T, Hemingway-Foday J, McClure EM, Koso-Thomas M, Derman RJ, Hoffman M, Bauserman M. Predictors of Plasmodium falciparum Infection in the First Trimester Among Nulliparous Women From Kenya, Zambia, and the Democratic Republic of the Congo. J Infect Dis. 2022 Jun 1;225(11):2002-2010. doi: 10.1093/infdis/jiab588. PMID 34888658
- [Background] Jafari-Guemouri S, Courtois L, Mama A, Rouas B, Neto Braga G, Accrombessi M, Massougbodji A, Ding XC, Tuikue Ndam N, Fievet N, Briand V. A Genotyping Study in Benin Comparing the Carriage of Plasmodium falciparum Infections Before Pregnancy and in Early Pregnancy: Story of a Persistent Infection. Clin Infect Dis. 2021 Jul 15;73(2):e355-e361. doi: 10.1093/cid/ciaa841. PMID 32569359
- [Background] Hounkonnou CPA, Briand V, Fievet N, Accrombessi M, Yovo E, Mama A, Sossou D, Vianou B, Massougbodji A, Ndam NT, Cot M, Cottrell G. Dynamics of Submicroscopic Plasmodium falciparum Infections Throughout Pregnancy: A Preconception Cohort Study in Benin. Clin Infect Dis. 2020 Jun 24;71(1):166-174. doi: 10.1093/cid/ciz748. PMID 32215629
- [Background] Tuikue Ndam N, Tornyigah B, Dossou AY, Escriou G, Nielsen MA, Salanti A, Issifou S, Massougbodji A, Chippaux JP, Deloron P. Persistent Plasmodium falciparum Infection in Women With an Intent to Become Pregnant as a Risk Factor for Pregnancy-associated Malaria. Clin Infect Dis. 2018 Nov 28;67(12):1890-1896. doi: 10.1093/cid/ciy380. PMID 29733338
- [Background] Briand V, Cottrell G, Tuike Ndam N, Martianez-Vendrell X, Vianou B, Mama A, Kouwaye B, Houze S, Bailly J, Gbaguidi E, Sossou D, Massougbodji A, Accrombessi M, Mayor A, Ding XC, Fievet N. Prevalence and clinical impact of malaria infections detected with a highly sensitive HRP2 rapid diagnostic test in Beninese pregnant women. Malar J. 2020 May 24;19(1):188. doi: 10.1186/s12936-020-03261-1. PMID 32448310
- [Background] Tagbor H, Cairns M, Bojang K, Coulibaly SO, Kayentao K, Williams J, Abubakar I, Akor F, Mohammed K, Bationo R, Dabira E, Soulama A, Djimde M, Guirou E, Awine T, Quaye S, Njie F, Ordi J, Doumbo O, Hodgson A, Oduro A, Meshnick S, Taylor S, Magnussen P, ter Kuile F, Woukeu A, Milligan P, Chandramohan D, Greenwood B. A Non-Inferiority, Individually Randomized Trial of Intermittent Screening and Treatment versus Intermittent Preventive Treatment in the Control of Malaria in Pregnancy. PLoS One. 2015 Aug 10;10(8):e0132247. doi: 10.1371/journal.pone.0132247. eCollection 2015. PMID 26258474
- [Background] Taylor SM, Madanitsa M, Thwai KL, Khairallah C, Kalilani-Phiri L, van Eijk AM, Mwapasa V, Ter Kuile FO, Meshnick SR. Minimal Impact by Antenatal Subpatent Plasmodium falciparum Infections on Delivery Outcomes in Malawian Women: A Cohort Study. J Infect Dis. 2017 Aug 1;216(3):296-304. doi: 10.1093/infdis/jix304. PMID 28658935
- [Background] Cottrell G, Moussiliou A, Luty AJ, Cot M, Fievet N, Massougbodji A, Deloron P, Tuikue Ndam N. Submicroscopic Plasmodium falciparum Infections Are Associated With Maternal Anemia, Premature Births, and Low Birth Weight. Clin Infect Dis. 2015 May 15;60(10):1481-8. doi: 10.1093/cid/civ122. Epub 2015 Feb 18. PMID 25694651
- [Background] Dorman EK, Shulman CE, Kingdom J, Bulmer JN, Mwendwa J, Peshu N, Marsh K. Impaired uteroplacental blood flow in pregnancies complicated by falciparum malaria. Ultrasound Obstet Gynecol. 2002 Feb;19(2):165-70. doi: 10.1046/j.0960-7692.2001.00545.x. PMID 11876809
- [Background] Umbers AJ, Stanisic DI, Ome M, Wangnapi R, Hanieh S, Unger HW, Robinson LJ, Lufele E, Baiwog F, Siba PM, King CL, Beeson JG, Mueller I, Aplin JD, Glazier JD, Rogerson SJ. Does malaria affect placental development? Evidence from in vitro models. PLoS One. 2013;8(1):e55269. doi: 10.1371/journal.pone.0055269. Epub 2013 Jan 31. PMID 23383132
- [Background] Conroy AL, Silver KL, Zhong K, Rennie M, Ward P, Sarma JV, Molyneux ME, Sled J, Fletcher JF, Rogerson S, Kain KC. Complement activation and the resulting placental vascular insufficiency drives fetal growth restriction associated with placental malaria. Cell Host Microbe. 2013 Feb 13;13(2):215-26. doi: 10.1016/j.chom.2013.01.010. PMID 23414761
- [Background] Elphinstone RE, Weckman AM, McDonald CR, Tran V, Zhong K, Madanitsa M, Kalilani-Phiri L, Khairallah C, Taylor SM, Meshnick SR, Mwapasa V, Ter Kuile FO, Conroy AL, Kain KC. Early malaria infection, dysregulation of angiogenesis, metabolism and inflammation across pregnancy, and risk of preterm birth in Malawi: A cohort study. PLoS Med. 2019 Oct 1;16(10):e1002914. doi: 10.1371/journal.pmed.1002914. eCollection 2019 Oct. PMID 31574087
- [Background] Moeller SL, Nyengaard JR, Larsen LG, Nielsen K, Bygbjerg IC, Msemo OA, Lusingu JPA, Minja DTR, Theander TG, Schmiegelow C. Malaria in Early Pregnancy and the Development of the Placental Vasculature. J Infect Dis. 2019 Sep 26;220(9):1425-1434. doi: 10.1093/infdis/jiy735. PMID 30590576
- [Background] Rijken MJ, Papageorghiou AT, Thiptharakun S, Kiricharoen S, Dwell SL, Wiladphaingern J, Pimanpanarak M, Kennedy SH, Nosten F, McGready R. Ultrasound evidence of early fetal growth restriction after maternal malaria infection. PLoS One. 2012;7(2):e31411. doi: 10.1371/journal.pone.0031411. Epub 2012 Feb 9. PMID 22347473
- [Background] Griffin JB, Lokomba V, Landis SH, Thorp JM Jr, Herring AH, Tshefu AK, Rogerson SJ, Meshnick SR. Plasmodium falciparum parasitaemia in the first half of pregnancy, uterine and umbilical artery blood flow, and foetal growth: a longitudinal Doppler ultrasound study. Malar J. 2012 Sep 10;11:319. doi: 10.1186/1475-2875-11-319. PMID 22963509
- [Background] Das S, Jang IK, Barney B, Peck R, Rek JC, Arinaitwe E, Adrama H, Murphy M, Imwong M, Ling CL, Proux S, Haohankhunnatham W, Rist M, Seilie AM, Hanron A, Daza G, Chang M, Nakamura T, Kalnoky M, Labarre P, Murphy SC, McCarthy JS, Nosten F, Greenhouse B, Allauzen S, Domingo GJ. Performance of a High-Sensitivity Rapid Diagnostic Test for Plasmodium falciparum Malaria in Asymptomatic Individuals from Uganda and Myanmar and Naive Human Challenge Infections. Am J Trop Med Hyg. 2017 Nov;97(5):1540-1550. doi: 10.4269/ajtmh.17-0245. Epub 2017 Aug 18. PMID 28820709
- [Background] Landier J, Haohankhunnatham W, Das S, Konghahong K, Christensen P, Raksuansak J, Phattharakokoedbun P, Kajeechiwa L, Thwin MM, Jang IK, Imwong M, Wiladphaingern J, Lwin KM, Ling C, Proux S, Domingo GJ, Delmas G, Nosten FH. Operational Performance of a Plasmodium falciparum Ultrasensitive Rapid Diagnostic Test for Detection of Asymptomatic Infections in Eastern Myanmar. J Clin Microbiol. 2018 Jul 26;56(8):e00565-18. doi: 10.1128/JCM.00565-18. Print 2018 Aug. PMID 29898998
- [Background] Slater HC, Ding XC, Knudson S, Bridges DJ, Moonga H, Saad NJ, De Smet M, Bennett A, Dittrich S, Slutsker L, Domingo GJ. Performance and utility of more highly sensitive malaria rapid diagnostic tests. BMC Infect Dis. 2022 Feb 4;22(1):121. doi: 10.1186/s12879-021-07023-5. PMID 35120441
- [Background] Vasquez AM, Velez G, Medina A, Serra-Casas E, Campillo A, Gonzalez IJ, Murphy SC, Seilie AM, Ding XC, Tobon Castano A. Evaluation of highly sensitive diagnostic tools for the detection of P. falciparum in pregnant women attending antenatal care visits in Colombia. BMC Pregnancy Childbirth. 2020 Jul 31;20(1):440. doi: 10.1186/s12884-020-03114-4. PMID 32736543
- [Background] Vasquez AM, Medina AC, Tobon-Castano A, Posada M, Velez GJ, Campillo A, Gonzalez IJ, Ding X. Performance of a highly sensitive rapid diagnostic test (HS-RDT) for detecting malaria in peripheral and placental blood samples from pregnant women in Colombia. PLoS One. 2018 Aug 2;13(8):e0201769. doi: 10.1371/journal.pone.0201769. eCollection 2018. PMID 30071004
- [Background] Unwin VT, Ahmed R, Noviyanti R, Puspitasari AM, Utami RAS, Trianty L, Lukito T, Syafruddin D, Poespoprodjo JR, Santana-Morales MA, Ter Kuile FO, Adams ER. Use of a highly-sensitive rapid diagnostic test to screen for malaria in pregnancy in Indonesia. Malar J. 2020 Jan 16;19(1):28. doi: 10.1186/s12936-020-3110-6. PMID 31948448
- [Background] Burger RJ, van Eijk AM, Bussink M, Hill J, Ter Kuile FO. Artemisinin-Based Combination Therapy Versus Quinine or Other Combinations for Treatment of Uncomplicated Plasmodium falciparum Malaria in the Second and Third Trimester of Pregnancy: A Systematic Review and Meta-Analysis. Open Forum Infect Dis. 2015 Nov 12;3(1):ofv170. doi: 10.1093/ofid/ofv170. eCollection 2016 Jan. PMID 26788543
- [Background] PREGACT Study Group; Pekyi D, Ampromfi AA, Tinto H, Traore-Coulibaly M, Tahita MC, Valea I, Mwapasa V, Kalilani-Phiri L, Kalanda G, Madanitsa M, Ravinetto R, Mutabingwa T, Gbekor P, Tagbor H, Antwi G, Menten J, De Crop M, Claeys Y, Schurmans C, Van Overmeir C, Thriemer K, Van Geertruyden JP, D'Alessandro U, Nambozi M, Mulenga M, Hachizovu S, Kabuya JB, Mulenga J. Four Artemisinin-Based Treatments in African Pregnant Women with Malaria. N Engl J Med. 2016 Mar 10;374(10):913-27. doi: 10.1056/NEJMoa1508606. PMID 26962727
- [Background] Kovacs SD, van Eijk AM, Sevene E, Dellicour S, Weiss NS, Emerson S, Steketee R, Ter Kuile FO, Stergachis A. The Safety of Artemisinin Derivatives for the Treatment of Malaria in the 2nd or 3rd Trimester of Pregnancy: A Systematic Review and Meta-Analysis. PLoS One. 2016 Nov 8;11(11):e0164963. doi: 10.1371/journal.pone.0164963. eCollection 2016. PMID 27824884
- [Background] Clark RL, White TE, A Clode S, Gaunt I, Winstanley P, Ward SA. Developmental toxicity of artesunate and an artesunate combination in the rat and rabbit. Birth Defects Res B Dev Reprod Toxicol. 2004 Dec;71(6):380-94. doi: 10.1002/bdrb.20027. PMID 15617018
- [Background] Clark RL, Lerman SA, Cox EM, Gristwood WE, White TE. Developmental toxicity of artesunate in the rat: comparison to other artemisinins, comparison of embryotoxicity and kinetics by oral and intravenous routes, and relationship to maternal reticulocyte count. Birth Defects Res B Dev Reprod Toxicol. 2008 Aug;83(4):397-406. doi: 10.1002/bdrb.20165. PMID 18702118
- [Background] Clark RL. Animal Embryotoxicity Studies of Key Non-Artemisinin Antimalarials and Use in Women in the First Trimester. Birth Defects Res. 2017 Aug 15;109(14):1075-1126. doi: 10.1002/bdr2.1035. Epub 2017 Jun 24. PMID 28646540
- [Background] Dellicour S, Sevene E, McGready R, Tinto H, Mosha D, Manyando C, Rulisa S, Desai M, Ouma P, Oneko M, Vala A, Ruperez M, Macete E, Menendez C, Nakanabo-Diallo S, Kazienga A, Valea I, Calip G, Augusto O, Genton B, Njunju EM, Moore KA, d'Alessandro U, Nosten F, Ter Kuile F, Stergachis A. First-trimester artemisinin derivatives and quinine treatments and the risk of adverse pregnancy outcomes in Africa and Asia: A meta-analysis of observational studies. PLoS Med. 2017 May 2;14(5):e1002290. doi: 10.1371/journal.pmed.1002290. eCollection 2017 May. PMID 28463996
- [Background] Ballard SB, Salinger A; MPHc; Arguin PM, Desai M, Tan KR. Updated CDC Recommendations for Using Artemether-Lumefantrine for the Treatment of Uncomplicated Malaria in Pregnant Women in the United States. MMWR Morb Mortal Wkly Rep. 2018 Apr 13;67(14):424-431. doi: 10.15585/mmwr.mm6714a4. PMID 29649190
- [Background] Kayentao K, Doumbo OK, Penali LK, Offianan AT, Bhatt KM, Kimani J, Tshefu AK, Kokolomami JH, Ramharter M, de Salazar PM, Tiono AB, Ouedraogo A, Bustos MD, Quicho F, Borghini-Fuhrer I, Duparc S, Shin CS, Fleckenstein L. Pyronaridine-artesunate granules versus artemether-lumefantrine crushed tablets in children with Plasmodium falciparum malaria: a randomized controlled trial. Malar J. 2012 Oct 31;11:364. doi: 10.1186/1475-2875-11-364. PMID 23113947
- [Background] Longo M, Pace S, Messina M, Ferraris L, Brughera M, Ubben D, Mazue G. Piperaquine phosphate: reproduction studies. Reprod Toxicol. 2012 Dec;34(4):584-97. doi: 10.1016/j.reprotox.2012.09.001. Epub 2012 Sep 19. PMID 23000234
- [Background] Batty KT, Moore BR, Stirling V, Ilett KF, Page-Sharp M, Shilkin KB, Mueller I, Karunajeewa HA, Davis TM. Toxicology and pharmacokinetics of piperaquine in mice. Toxicology. 2008 Jul 10;249(1):55-61. doi: 10.1016/j.tox.2008.04.004. Epub 2008 Apr 16. PMID 18502018
- [Background] Bretscher MT, Dahal P, Griffin J, Stepniewska K, Bassat Q, Baudin E, D'Alessandro U, Djimde AA, Dorsey G, Espie E, Fofana B, Gonzalez R, Juma E, Karema C, Lasry E, Lell B, Lima N, Menendez C, Mombo-Ngoma G, Moreira C, Nikiema F, Ouedraogo JB, Staedke SG, Tinto H, Valea I, Yeka A, Ghani AC, Guerin PJ, Okell LC. The duration of chemoprophylaxis against malaria after treatment with artesunate-amodiaquine and artemether-lumefantrine and the effects of pfmdr1 86Y and pfcrt 76T: a meta-analysis of individual patient data. BMC Med. 2020 Feb 25;18(1):47. doi: 10.1186/s12916-020-1494-3. PMID 32098634
- [Background] Clark RL, Youreneff M, DeLise AM. Developmental toxicity studies of lumefantrine and artemether in rats and rabbits. Birth Defects Res B Dev Reprod Toxicol. 2016 Dec;107(6):243-257. doi: 10.1002/bdrb.21189. PMID 28032463
- [Background] Manyando C, Mkandawire R, Puma L, Sinkala M, Mpabalwani E, Njunju E, Gomes M, Ribeiro I, Walter V, Virtanen M, Schlienger R, Cousin M, Chipimo M, Sullivan FM. Safety of artemether-lumefantrine in pregnant women with malaria: results of a prospective cohort study in Zambia. Malar J. 2010 Sep 1;9:249. doi: 10.1186/1475-2875-9-249. PMID 20809964
- [Background] Rulisa S, Kaligirwa N, Agaba S, Karema C, Mens PF, de Vries PJ. Pharmacovigilance of artemether-lumefantrine in pregnant women followed until delivery in Rwanda. Malar J. 2012 Jul 6;11:225. doi: 10.1186/1475-2875-11-225. PMID 22770264
- [Background] Mosha D, Mazuguni F, Mrema S, Sevene E, Abdulla S, Genton B. Safety of artemether-lumefantrine exposure in first trimester of pregnancy: an observational cohort. Malar J. 2014 May 27;13:197. doi: 10.1186/1475-2875-13-197. PMID 24884890
- [Background] Dellicour S, Desai M, Aol G, Oneko M, Ouma P, Bigogo G, Burton DC, Breiman RF, Hamel MJ, Slutsker L, Feikin D, Kariuki S, Odhiambo F, Pandit J, Laserson KF, Calip G, Stergachis A, ter Kuile FO. Risks of miscarriage and inadvertent exposure to artemisinin derivatives in the first trimester of pregnancy: a prospective cohort study in western Kenya. Malar J. 2015 Nov 18;14:461. doi: 10.1186/s12936-015-0950-6. PMID 26581434
- [Background] Augusto O, Stergachis A, Dellicour S, Tinto H, Vala A, Ruperez M, Macete E, Nakanabo-Diallo S, Kazienga A, Valea I, d'Alessandro U, Ter Kuile FO, Calip GS, Ouma P, Desai M, Sevene E. First trimester use of artemisinin-based combination therapy and the risk of low birth weight and small for gestational age. Malar J. 2020 Apr 8;19(1):144. doi: 10.1186/s12936-020-03210-y. PMID 32268901
- [Background] Walker PG, ter Kuile FO, Garske T, Menendez C, Ghani AC. Estimated risk of placental infection and low birthweight attributable to Plasmodium falciparum malaria in Africa in 2010: a modelling study. Lancet Glob Health. 2014 Aug;2(8):e460-7. doi: 10.1016/S2214-109X(14)70256-6. Epub 2014 Jul 23. PMID 25103519
- [Background] Kapito-Tembo A, Meshnick SR, van Hensbroek MB, Phiri K, Fitzgerald M, Mwapasa V. Marked reduction in prevalence of malaria parasitemia and anemia in HIV-infected pregnant women taking cotrimoxazole with or without sulfadoxine-pyrimethamine intermittent preventive therapy during pregnancy in Malawi. J Infect Dis. 2011 Feb 15;203(4):464-72. doi: 10.1093/infdis/jiq072. Epub 2011 Jan 7. PMID 21216867
- [Background] ACOG committee opinion no. 561: Nonmedically indicated early-term deliveries. Obstet Gynecol. 2013 Apr;121(4):911-915. doi: 10.1097/01.AOG.0000428649.57622.a7. PMID 23635710
- [Background] Hoffman MK, Goudar SS, Kodkany BS, Metgud M, Somannavar M, Okitawutshu J, Lokangaka A, Tshefu A, Bose CL, Mwapule A, Mwenechanya M, Chomba E, Carlo WA, Chicuy J, Figueroa L, Garces A, Krebs NF, Jessani S, Zehra F, Saleem S, Goldenberg RL, Kurhe K, Das P, Patel A, Hibberd PL, Achieng E, Nyongesa P, Esamai F, Liechty EA, Goco N, Hemingway-Foday J, Moore J, Nolen TL, McClure EM, Koso-Thomas M, Miodovnik M, Silver R, Derman RJ; ASPIRIN Study Group. Low-dose aspirin for the prevention of preterm delivery in nulliparous women with a singleton pregnancy (ASPIRIN): a randomised, double-blind, placebo-controlled trial. Lancet. 2020 Jan 25;395(10220):285-293. doi: 10.1016/S0140-6736(19)32973-3. PMID 31982074
- [Background] Landis SH, Lokomba V, Ananth CV, Atibu J, Ryder RW, Hartmann KE, Thorp JM, Tshefu A, Meshnick SR. Impact of maternal malaria and under-nutrition on intrauterine growth restriction: a prospective ultrasound study in Democratic Republic of Congo. Epidemiol Infect. 2009 Feb;137(2):294-304. doi: 10.1017/S0950268808000915. Epub 2008 Jun 30. PMID 18588723
- See also: Organization WH. Every Newborn: an action plan to end preventable deaths. — http://www.healthynewbornnetwork.org/hnn-content/uploads/Every_Newborn_Action_Plan-ENGLISH_updated_July2014.pdf
- See also: WHO. Recommendations on intermittent screening and treatment in pregnancy and the safety of ACTs in the first trimester. — http://apps.who.int/iris/handle/10665/338496